CLINICAL TRIAL: NCT01913444
Title: Pharmacokinetics of Recombinant Antithrombin III in Neonates Undergoing Extracorporeal Membrane Oxygenation
Brief Title: Pharmacokinetic Study of Recombinant AT III in Neonates Undergoing ECMO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll patients into study.
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Philippe Samuel Friedlich, M.D, MD, MS Epi, MBA, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-12-00147
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Neonates on ECMO
Keywords: Recombinant Antithrombin; ATryn; Pharmacokinetics; ECMO; Neonates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant Antithrombin Infusion (Experimental): The initial loading dose and maintenance continuous infusion will be calculated according to the following equations which are based on the patient's baseline AT activity level prior to ECMO. Loading dose(IU)=(100-baseline AT activity)/2.3 x Wt(kg). Maintenance Dose(IU/hour)=(100-baseline AT activity)/10.2 x Wt(kg). The loading dose will be administered as a 15-minute IV infusion once the patient is on ECMO. This will be followed by the maintenance continuous infusion. AT levels will be checked 2hours after the initiation of treatment. For AT levels that are <80% or >100%, the infusion rate will be increased or decreased, respectively, by 30% and a follow-up level will be checked 2hours after the adjustment. If the AT level is within goal range (80-100%), follow-up AT levels will be checked every 6hours unless dose adjustments are made. Once the patient is off ECMO, the continuous infusion will be discontinued and AT levels will no longer be checked.
  Interventions: Drug: Recombinant Antithrombin

INTERVENTIONS:
Drug: Recombinant Antithrombin
  Other Names: ATryn

SUMMARY:
Maintenance of adequate anticoagulation or blood thinning is of critical importance when patients are placed on extracorporeal life support, such as extracorporeal membrane oxygenation (ECMO). During ECMO, a patient's entire blood volume is constantly exposed to the artificial surfaces of the ECMO circuit. This exposure activates the clotting cascade, and not only is the circuit at risk for clot formation, but the patient is also at risk for clotting within the body. Hence anticoagulation is vital in allowing the ECMO circuit to support a patient for an extended period of time. Anticoagulation on ECMO is achieved primarily by the use of a blood thinning agent called heparin. Heparin's main mechanism of action is to activate an enzyme called antithrombin III (AT III). AT III deficiency has been shown to be a common finding in pediatric patients requiring ECMO. This deficiency may then result in ineffective blood thinning by heparin. The purpose of this study is to determine how a neonate on ECMO, processes and eliminates a medication called ATryn® from their body. ATryn® is a form ATIII that is made from goat's milk. This will ultimately aid in establishing standardized dosing for the use of ATryn® in this patient population.

DETAILED DESCRIPTION:
Maintenance of adequate anticoagulation is of critical importance when patients are placed on extracorporeal life support, such as ECMO. During ECMO, a patient's entire blood volume is constantly exposed to the artificial surfaces of the ECMO circuit. This exposure activates the clotting cascade, and not only is the circuit at risk for clot formation, but the patient is also at risk for thromboembolic events. Hence anticoagulation is vital in allowing the ECMO circuit to support a patient's entire cardiopulmonary system for an extended period of time. Anticoagulation on ECMO is achieved primarily by the use of a heparin continuous infusion. Heparin's main mechanism of action is to bind to and activate an enzyme called antithrombin III (AT III). AT III is the principal inhibitor of the blood coagulation serine proteases - Thrombin and Factor Xa. In the presence of, and when bound to heparin, the inhibitory activity of AT III is greatly enhanced. AT III deficiency has been shown to be a common finding in pediatric patients requiring ECMO. Our center has reported that most neonatal patients requiring ECMO also have a significant degree of ATIII deficiency prior to, and during ECMO bypass. This deficiency may lead to challenges in achieving adequate anticoagulation while on ECMO. For this reason, our institution already supplements antithrombin during pre-ECMO circuit priming and for maintaining AT III levels above 70% during the entire length of ECMO support. Optimizing AT III levels may then improve anticoagulation while on ECMO. This study aims to determine the pharmacokinetics of recombinant antithrombin (ATryn®) supplementation. To date, the use of ATryn® has primarily been studied in adults. There is no published data to date, and no current studies on the pharmacokinetics of antithrombin III in neonates, and hence no published data on the pharmacokinetics of antithrombin III in the neonatal ECMO population. Since the use of antithrombin III in the neonatal ECMO patient population has not been thoroughly studied, the use of antithrombin III supplementation varies greatly among different neonatal intensive care units. Therefore, studies that aim at determining the pharmacokinetics of antithrombin III, particularly in ECMO patients, are important because of the lack of data and published studies in this patient population. By determining the pharmacokinetics of ATryn® in our neonatal ECMO patient population, we will aid in establishing standardized dosing and administration protocols for the supplementation of antithrombin in this specific patient population.

Summary of Risks and Benefits: ATryn® is FDA approved for use in the prevention of peri-operative and peri-partum thromboembolic events in hereditary antithrombin III deficient patients. ATryn® is a transgenically produced recombinant antithrombin concentrate from goat milk that is preservative free. It has an identical amino acid structure with minor glycosylation differences to endogenous human AT IIII. When assayed in the presence of excess heparin, the potency and efficacy of ATryn® is not different from that of plasma-derived AT III concentrates.5 ATryn® is administered as a continuous intravenous infusion, with weight-adjusted loading and maintenance dosing regimens as recommended by the medication's package insert. As dosing is specific to a patient's weight, this theoretically minimizes the risk for overdosing. In addition, as dosing is administered as a continuous infusion that is titrated to maintain stable AT III levels, there is the additional potential for less fluctuations in a patient's AT III levels. Not only will anticoagulation be optimized throughout the duration of ECMO support, but theoretically there may be a decreased need for, or less fluctuations in a patient's heparin requirements. This may furthermore minimize the risk for thromboembolic events within the ECMO circuit and the patient. Additionally, ATryn® is preservative free and because it is a recombinant product, it should be free from the risk of viral infection or prion transmission.

ELIGIBILITY:
Inclusion Criteria:

* Neonates requiring ECMO
* Must be < or = to 30 days of age
* Must be > or = to 37weeks corrected gestational age

Exclusion Criteria:

* Older than or = to 31 days of age
* Preterm neonates < 37weeks corrected gestational age
* Previously diagnosed hereditary coagulopathy or hemorrhagic disorder in the family
* Prior to recent anticoagulation use
* Known or suspected genetic or terminal disorder
* Known family history of hypersensitivity to goat's milk or goat milk products

Ages: 1 Minute to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Antithrombin III Level | Every 6 hours until steady state within first 72 hours on ECMO
  ATIII levels will be checked at a minimum of every 6 hours throughout a patient's ECMO course. However, should dose adjustments be made to the ATryn infusion rate, ATIII levels will be checked 2hours after each dose adjustment. Once the ATIII level is again within goal range, ATIII levels will resume to being checked every 6hours.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe S Friedlich, MD, MS Epi, MBA, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Niebler RA, Christensen M, Berens R, Wellner H, Mikhailov T, Tweddell JS. Antithrombin replacement during extracorporeal membrane oxygenation. Artif Organs. 2011 Nov;35(11):1024-8. doi: 10.1111/j.1525-1594.2011.01384.x. PMID 22097980
- [Background] Agati S, Ciccarello G, Salvo D, Turla G, Undar A, Mignosa C. Use of a novel anticoagulation strategy during ECMO in a pediatric population: single-center experience. ASAIO J. 2006 Sep-Oct;52(5):513-6. doi: 10.1097/01.mat.0000242596.92625.a0. PMID 16966848
- [Background] Sievert A, Uber W, Laws S, Cochran J. Improvement in long-term ECMO by detailed monitoring of anticoagulation: a case report. Perfusion. 2011 Jan;26(1):59-64. doi: 10.1177/0267659110385513. Epub 2010 Nov 5. PMID 21057061
- [Background] Konkle BA, Bauer KA, Weinstein R, Greist A, Holmes HE, Bonfiglio J. Use of recombinant human antithrombin in patients with congenital antithrombin deficiency undergoing surgical procedures. Transfusion. 2003 Mar;43(3):390-4. doi: 10.1046/j.1537-2995.2003.00315.x. PMID 12675726